CLINICAL TRIAL: NCT06631742
Title: The Effect of an Exergaming Intervention on Physical Activity and Sleep in People With Major Neurocognitive Disorders Living in Long-term Care Facilities: a Pilot Randomized Controlled Trial.
Brief Title: Exergaming Revolution in Dementia
Acronym: GameDementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Eling de Bruin, Prof. Dr. Eling de Bruin, Eastern Switzerland University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-00113.
Record Dates: First submitted 2024-09-10; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Major Neurocognitive Disorder; Alzheimer Disease; Parkinson Disease; Lewy Body Dementia; Mixed Dementias
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Lewy Body Disease; Mixed Dementias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): Individual active dance game training on Dividat Senso
  Interventions: Other: Exergaming on Dividat Senso
- Usual Care (Other): Customised care and support as required
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exergaming on Dividat Senso — The active dance video game is played with the Dividat Senso (Dividat | Senso: cognitive-motor training). It consists of a dance disc with four arrows (up, down, left, right), and the game is played on a large screen (which is connected to the PC). The screen indicates which arrow the person should step on, thus controlling the game through body movements. The games give the person feedback in the form of auditory, visual, and somatosensory stimuli.
  Arms: Exergaming
Other: Usual Care — Standardised care with meal service, individual activities (e.g. hiking group, walking group, exercise group, handicrafts, gardening group, singing, painting or lunch) and customized care and support as required.
  Arms: Usual Care

SUMMARY:
This pilot randomized controlled trial evaluates the effect of a 12 weeks exergaming training in people with major neurocognitive disorders (MNCD) living in long-term care facilities.

DETAILED DESCRIPTION:
Background: Major neurocogntivie disorders (MNCD) are categorised as public health priority by the World Health Organisation. To date, there are no disease-modifying treatments that can cure MNCD or effectively halt its progression. However, lifestyle changes that increase physical activity and/or reduce vascular risk factors are effective in protecting against brain atrophy and cognitive decline. Therefore, it has been suggested to focus on non-pharmacological therapies that target people's lifestyle, such as multimodal treatment strategies that encompass multiple domains, including physical exercise and cognitive stimulation. Exergames which combine exercise with feedback on performance, fun, relaxation and socialising, are promising for older people.

The goal of this pilot randomized controlled trial is to evaluate the effect of an exergaming intervention in people with MNCD. The main questions it aims to answer are:

* How does an exergaming intervention effects gait speed, cognitive and motor functions as well as depressive symptoms and quality of life in residents of a long-term care facilities.
* How does an exergaming intervention effects physical activity and sleep in residents of a long-term care facilities.

Methods: Investigators plan to include 48 participants living in long-term care facilities. Participants will participate in a 12 weeks active dance video game (3x 15minute per week) or will get care as usual. The Short Physical Perfomance Battery (SPPB), The Montréal Cognitive Assessment (MoCA), Neuropsychiatric Inventory (NPI), Cornell Scale for Depression in Dementia (CSDD), Quality of Life in Alzheimer's (QoL-AD), Katz activities of daily living (Katz-ADL), Geriatric Sleep Questionnaire (GSQ-6), number's of falls in the last 12 weeks, physical activity and sleep parameters of the motions sensor GENEactiv and sleep parameters of the contacless sensorbox Sleepiz are measured at baseline and post intervention.

For all outcomes, descriptive statistics will be computed first. Normality distribution of data will be checked using the Shapiro-Wilk test and Q-Q-plots. The assumptions of homogeneity of variance and of sphericity will be checked using Levene's test and Mauchly's test, respectively. In case all assumptions are met, a two-way analysis of covariance (ANCOVA) will be computed for all primary and secondary outcomes with the pre-test as covariate for the predicting group factor and the posttest as outcome variable. Therefore, the outcome is the differences of the pre- and post-test with the baseline as the influencing variable. In case not all assumptions for ANCOVA are met, Quade non-parametric tests will be used. The level of significance will be set to p ≤ 0.05 (two-sided).

ELIGIBILITY:
Inclusion Criteria:

* Neurocognitive disorder based on Alzheimer's Disease, Parkinson's disease, Lewy body dementia or Mixed dementia according to the criteria of the American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5)
* Mini-Mental-Status-Examination (MMSE) Score of ≥5 and ≤26 out of e maximum of 30

Exclusion Criteria:

* MMSE <5
* Unstable cardiovascular condition or other medical condition that does not allow for safe participation according to the recommendations of the American College of Sports Medicine
* Planned transfer to another facility within the next 3 months
* Acute behavioural problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline
  The SPPB is developed by the National Institute of Aging (NIA). It is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (> 65 years of age). The test battery consists of three physical tasks (walking, sit-to-stand and balance) to assess functional mobility. The test will be performed according to standardised procedure. The maximal total score is 12 and higher total scores indicate a better lower extremity functioning.
Short Phyiscal Performance Battery | after 12 weeks
  The SPPB is developed by the National Institute of Aging (NIA). It is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (> 65 years of age). The test battery consists of three physical tasks (walking, sit-to-stand and balance) to assess functional mobility. The test will be performed according to standardised procedure. The maximal total score is 12 and higher total scores indicate a better lower extremity functioning.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Baseline, after 12 weeks
  The MoCA is a objective instrument, which is designed for milder forms of major neurocognitive disorders, contains 12 items to assess seven cognitive domains: memory, language, executive functions, visuospatial skills, attention, concentration, abstraction, calculation, and orientation. The maximal total score is 30 and higher total score indicate less cognitive impairment. A cut-off score of 26 signifies mild cognitive impairment.
Neuropsychiatric Inventory Questionnaire | Baseline, after 12 weeks
  The NPI-Q assesses psychopathological problems and is designed to be a self-administered questionnaire completed by caregivers. The questionnaire screening symptom severity and caregiver distress of the following 12 domains: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviour, night-time behaviour disturbance, and appetite and eating abnormalities. The symptom severity scale ranging from 1 to 3. The caregiver distress scale ranging from 0 to 5. The NPI total score is calculated by multiplying the frequency and severity rates per domain and adding them up. The total score ranges from 0 to 144, with higher score indicating hight severity and higher distress.
Cornell Scale for Depression in Dementia | Baseline, after 12 weeks
  The observation based CSDD, in the form of an interview with the caregiver assesses symptoms of depression. The CSDD consists of 19 items and each one is scored on a 3-point scale ranging from 0 to 2. Items are clustered into five categories: mood, behavioural disturbance, physical signs, cyclic functions, and ideational disturbance. The maximum score is 38, and higher score indicating more depressive symptoms.
Quality of Life in Alzheimer's | Baseline, after 12 weeks
  The QOL-AD is a brief, 13-item which assesses individual's relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality. It is designed to acquire a rating of the patient's Quality of Life from both the patient and the caregiver. It uses simple and straightforward language and responses and includes assessments of the caregivers complete the measure as a questionnaire about their patients' QOL, while patients complete it in interview format about their own QOL. The 13 items are rated on a four-point Likert scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52. The sum of all items; patient and caregiver reports can be evaluated separately and/or combined into a single score if desired.
Katz ADL | Baseline, after 12 weeks
  The interviewer-administered Katz ADL Index assesses participants' function in terms of level of independence or dependence when performing certain daily living activities. It consists of six items: bathing, dressing, transfers, toileting, continence, and feeding. Each item is scored 0 (dependence) or 1 (independence) with a maximum score of 6, which indicates more independence.
Geriatric Sleep Questionnaire | Baseline, after 12 weeks
  Self-reported Questionnaire assesses overall sleep quality. Item score are summed up with the maximal total score of 30. Higher score indicate poorer sleep quality.
Numbers of falls in the last 12 weeks | Baseline, after 12 weeks
  Numbers of Falls during 12 weeks prior to baseline and during the 12 weeks to follow up according to the patient's medical record will be assessed.
Motion Sensor GENEactiv | Basline, after 12 weeks
  GENEActiv is a lightweight and waterproof medical device that delivers continuous recording of high-resolution acceleration that allows a person's daily activities to be classified, second by second, in terms of the time spent lying, sitting, standing, stepping and sleep parameters such as total sleep time, sleep efficiency and body temperature (e.g., circadian rhythm).
Contactless Sensorbox Sleepiz | Baseline, after 12 weeks
  Radar-based contactless technology measuring body position and respiratory rate.

CONTACTS AND LOCATIONS:
Overall Officials: Eling de Bruin, Prof. Dr., Principal Investigator — Eastern Swiss University of Applied Sciences
Locations (1):
- Sonnweid AG, Wetzikon, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Bellettiere J, Lamonte MJ, Unkart J, Liles S, Laddu-Patel D, Manson JE, Banack H, Seguin-Fowler R, Chavez P, Tinker LF, Wallace RB, LaCroix AZ. Short Physical Performance Battery and Incident Cardiovascular Events Among Older Women. J Am Heart Assoc. 2020 Jul 21;9(14):e016845. doi: 10.1161/JAHA.120.016845. Epub 2020 Jul 14. PMID 32662311
- [Result] Cassidy B, Arena S. The Short Physical Performance Battery as a Predictor of Functional Decline. Home Healthc Now. 2022 May-Jun 01;40(3):168-169. doi: 10.1097/NHH.0000000000001070. No abstract available. PMID 35510973
- [Result] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Result] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Result] Lindbergh CA, Dishman RK, Miller LS. Functional Disability in Mild Cognitive Impairment: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2016 Jun;26(2):129-59. doi: 10.1007/s11065-016-9321-5. Epub 2016 Jul 8. PMID 27393566
- [Result] Sanford AM. Mild Cognitive Impairment. Clin Geriatr Med. 2017 Aug;33(3):325-337. doi: 10.1016/j.cger.2017.02.005. Epub 2017 May 17. PMID 28689566
- [Result] Tisher A, Salardini A. A Comprehensive Update on Treatment of Dementia. Semin Neurol. 2019 Apr;39(2):167-178. doi: 10.1055/s-0039-1683408. Epub 2019 Mar 29. PMID 30925610
- [Result] Erickson KI, Raji CA, Lopez OL, Becker JT, Rosano C, Newman AB, Gach HM, Thompson PM, Ho AJ, Kuller LH. Physical activity predicts gray matter volume in late adulthood: the Cardiovascular Health Study. Neurology. 2010 Oct 19;75(16):1415-22. doi: 10.1212/WNL.0b013e3181f88359. Epub 2010 Oct 13. PMID 20944075
- [Result] Guure CB, Ibrahim NA, Adam MB, Said SM. Impact of Physical Activity on Cognitive Decline, Dementia, and Its Subtypes: Meta-Analysis of Prospective Studies. Biomed Res Int. 2017;2017:9016924. doi: 10.1155/2017/9016924. Epub 2017 Feb 7. PMID 28271072
- [Result] Vancampfort D, Solmi M, Firth J, Vandenbulcke M, Stubbs B. The Impact of Pharmacologic and Nonpharmacologic Interventions to Improve Physical Health Outcomes in People With Dementia: A Meta-Review of Meta-Analyses of Randomized Controlled Trials. J Am Med Dir Assoc. 2020 Oct;21(10):1410-1414.e2. doi: 10.1016/j.jamda.2020.01.010. Epub 2020 Feb 19. PMID 32085951
- [Result] Ahlskog JE, Geda YE, Graff-Radford NR, Petersen RC. Physical exercise as a preventive or disease-modifying treatment of dementia and brain aging. Mayo Clin Proc. 2011 Sep;86(9):876-84. doi: 10.4065/mcp.2011.0252. PMID 21878600
- [Result] Dimitrov DM, Rumrill PD Jr. Pretest-posttest designs and measurement of change. Work. 2003;20(2):159-65. PMID 12671209